CLINICAL TRIAL: NCT04459949
Title: Comparative Study of Sharkskin Versus Grieshaber Forceps During ILM Peeling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, MidAtlantic Retina, Principal Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #2020-91
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Epiretinal Membrane; Macular Holes
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sharkskin Arm (Active Comparator)
  Interventions: Device: Sharkskin
- Grieshaber Arm (Placebo Comparator)
  Interventions: Device: Grieshaber

INTERVENTIONS:
Device: Sharkskin — Use of Sharkskin ILM forceps
  Arms: Sharkskin Arm
Device: Grieshaber — Use of Grieshaber ILM forceps
  Arms: Grieshaber Arm

SUMMARY:
The purpose of this study is to compare the performance and anatomic outcomes of the Sharkskin internal limiting membrane (ILM) forceps and the Grieshaber ILM forceps in macular surgery.

Peeling of the ILM is a difficult aspect of vitreoretinal surgery and often daunting task from a vitreoretinal fellow's perspective. The hypothesis is that the newer Sharkskin forceps have a larger platform and micro-abrasions along the forcep surface to increase grasping ability and potentially limit trauma to the retina surface compared to the Grieshaber forceps. This project may also serve as an education tool for fellows learning the basics of ILM peeling.

ELIGIBILITY:
Inclusion Criteria:

* Macular pathology

Exclusion Criteria:

* No prior vitreoretinal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-06 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Surgical time | During surgery

SECONDARY OUTCOMES:
Ease of peeling - surgeon | During surgery
  Use of standardized questionnaire to the surgeon.
Ease of peeling - masked grader | Through study completion, up to one year
  Use of standardized questionnaire to the masked grader.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Starr MR, Hinkle JC, Patel LG, Ammar MJ, Soares RR, Patel SN, Cohen MN, Hsu J, Yonekawa Y, Ho AC, Regillo CD, Gupta OP. RANDOMIZED TRIAL COMPARING MICROSERRATED VERSUS CONVENTIONAL INTERNAL LIMITING MEMBRANE FORCEPS FOR INTERNAL LIMITING MEMBRANE PEELING. Retina. 2024 Aug 1;44(8):1323-1328. doi: 10.1097/IAE.0000000000004138. PMID 39047125